CLINICAL TRIAL: NCT06657118
Title: Ultrasound Guided Versus Conventional Arthrocentesis in Treatment of Temporomandibular Joint Internal Derangement: A Randomized Clinical Trial
Brief Title: Ultrasound Guided Versus Conventional Arthrocentesis in Treatment of Temporomandibular Joint Internal Derangement.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samiha Abdelsalam Abdelaziz Abdelaziz (Other)
Responsible Party: Sponsor-Investigator, Samiha Abdelsalam Abdelaziz Abdelaziz, Principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US guided arthrocentesis
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Internal Derangement of the Tempromandibular Joint

STUDY DESIGN:
Intervention Model Description: A randomized control trial, parallel group, allocation ratio 1:1 Framework equivalence
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional arthrocentesis (Active Comparator): * Scrubbing and draping of the patient will be carried out in a standard fashion using betadine surgical scrub.
  * Head turned to the affected side.
  * External auditory meatus will be blocked with a cotton plug.
  * A line will be drawn from tragus of the ear to the outer canthus of the eye with ink.
  * Double needled canula is inserted into superior compartment of the joint space 2mm below and 10 mm ahead of mid-tragal end of Holmund Hellsing's line.
  Intra-operative procedures - continued in both groups:
  * Lavage is performed with 100 ml of saline solution.
  * 1 ml of Hyaluronic acid is injected into the superior joint space.
  * Puncture point is covered with sterile dressing for 24 hours
  Interventions: Procedure: Conventional anatomically guided arthrocentesis of tempromandibular joint
- Ultrasound guided arthrocentesis (Active Comparator): Scrubbing and draping of the patient will be carried out in a standard fashion using betadine surgical scrub.
  * Head turned to the affected side.
  * External auditory meatus will be blocked with a cotton plug.
  * Transducer is placed over TMJ, parallel to the long axis of mandibular ramus. • Transducer is tilted until the optimal visualization is obtained.
  * Disc is visualized as a thin homogenous, hypo-to-iso-echoic band lying adjacent to the inferior relation. The bony landmarks of the mandibular condyle and the articular eminence are visualized as hyperdense lines.
  * Superior joint space located between the disc and articular eminence is the targeted point of the needle.
  Intra-operative procedures - continued in both groups:
  * Lavage is performed with 100 ml of saline solution.
  * 1 ml of Hyaluronic acid is injected into the superior joint space.
  * Puncture point is covered with sterile dressing for 24 hours
  Interventions: Procedure: Ultrasound guided arthrocentesis of tempromandibular joint

INTERVENTIONS:
Procedure: Ultrasound guided arthrocentesis of tempromandibular joint — * Scrubbing and draping of the patient will be carried out in a standard fashion using betadine surgical scrub.
  * Head turned to the affected side. • External auditory meatus will be blocked with a cotton plug.
  * Transducer is placed over TMJ, parallel to the long axis of mandibular ramus. • Transducer is tilted until the optimal visualization is obtained.
  * Disc is visualized as a thin homogenous, hypo-to-iso-echoic band lying adjacent to the inferior relation. The bony landmarks of the mandibular condyle and the articular eminence are visualized as hyperdense lines.
  * Superior joint space located between the disc and articular eminence is the targeted point of the needle.
  Intra-operative procedures - continued in both groups:
  * Lavage is performed with 100 ml of saline solution.
  * 1 ml of Hyaluronic acid is injected into the superior joint space.
  * Puncture point is covered with sterile dressing for 24 hours
  Arms: Ultrasound guided arthrocentesis
Procedure: Conventional anatomically guided arthrocentesis of tempromandibular joint — * Scrubbing and draping of the patient will be carried out in a standard fashion using betadine surgical scrub.
  * Head turned to the affected side. • External auditory meatus will be blocked with a cotton plug.
  * A line will be drawn from tragus of the ear to the outer canthus of the eye with ink.
  * Double needled canula is inserted into superior compartment of the joint space 2mm below and 10 mm ahead of mid-tragal end of Holmund Hellsing's line.
  Intra-operative procedures - continued in both groups:
  * Lavage is performed with 100 ml of saline solution.
  * 1 ml of Hyaluronic acid is injected into the superior joint space.
  * Puncture point is covered with sterile dressing for 24 hours
  Arms: Conventional arthrocentesis

SUMMARY:
The use of Ultrasound as a guide in arthrocentesis of tempromandibular joint versus conventional anatomically guided arthrocentesis in treatment of temporomandibular joint internal derangement: A randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 16 to 45 years of age having temporomandibular joint internal derangement.
* Patients free from any systemic conditions and bone metabolic diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.
* ASA 1-2 patients with no contraindications for GA
* Patients who did not respond to conservative treatment.

Exclusion Criteria:

* Patient with uncontrolled systemic diseases precluding administration of general anesthesia.
* Handicaps and special needs patients.
* Prisoners.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maximum mouth opening | Patients will be evaluated after 2 weeks from operation and every 2 weeks thereafter for the next 3 months.
  Maximum mouth opening of the patient will be measured in Millimetre (mm) using a ruler
Joint pain | Patients will be evaluated after 2 weeks from operation and every 2 weeks thereafter for the next 3 months.
  Joint pain: Will be measured by visual analogue scale (VAS) of 10 units according to pre-determined reference values: 0 No pain. 1-2 Faint pain. 3-4 Mild pain 5-6 Moderate pain. 7-8 Severe pain. 9-10 Excruciating pain.

SECONDARY OUTCOMES:
Operation time | Once during every procedure
  Operation time will be measured using stopwatch and recorded in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Moutaed, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
share it with other researchers websites if it is possible

REFERENCES:
- [Background] Dong XY, He S, Zhu L, Dong TY, Pan SS, Tang LJ, Zhu ZF. The diagnostic value of high-resolution ultrasonography for the detection of anterior disc displacement of the temporomandibular joint: a meta-analysis employing the HSROC statistical model. Int J Oral Maxillofac Surg. 2015 Jul;44(7):852-8. doi: 10.1016/j.ijom.2015.01.012. Epub 2015 Feb 20. PMID 25702588
- [Background] Maranini B, Ciancio G, Mandrioli S, Galie M, Govoni M. The Role of Ultrasound in Temporomandibular Joint Disorders: An Update and Future Perspectives. Front Med (Lausanne). 2022 Jun 20;9:926573. doi: 10.3389/fmed.2022.926573. eCollection 2022. PMID 35795636
- [Background] Poveda Roda R, Diaz Fernandez JM, Hernandez Bazan S, Jimenez Soriano Y, Margaix M, Sarrion G. A review of temporomandibular joint disease (TMJD). Part II: Clinical and radiological semiology. Morbidity processes. Med Oral Patol Oral Cir Bucal. 2008 Feb 1;13(2):E102-9. PMID 18223525
- [Background] Champs B, Corre P, Hamel A, Laffite CD, Le Goff B. US-guided temporomandibular joint injection: Validation of an in-plane longitudinal approach. J Stomatol Oral Maxillofac Surg. 2019 Feb;120(1):67-70. doi: 10.1016/j.jormas.2018.10.008. Epub 2018 Nov 6. PMID 30412740
- [Background] Bhargava D, Thomas S, Pawar P, Jain M, Pathak P. Ultrasound-guided arthrocentesis using single-puncture, double-lumen, single-barrel needle for patients with temporomandibular joint acute closed lock internal derangement. Oral Maxillofac Surg. 2019 Jun;23(2):159-165. doi: 10.1007/s10006-019-00753-6. Epub 2019 Mar 28. PMID 30923970
- [Background] Azlag Pekince K, Caglayan F, Pekince A. The efficacy and limitations of USI for diagnosing TMJ internal derangements. Oral Radiol. 2020 Jan;36(1):32-39. doi: 10.1007/s11282-019-00376-3. Epub 2019 Feb 4. PMID 30719601